CLINICAL TRIAL: NCT04035161
Title: Evaluation of the Antimicrobial Effectiveness of CHG/IPA in Healthy Volunteers
Brief Title: Evaluation of the Antimicrobial Effectiveness of CHG/IPA
Status: Completed | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MPS-17IPVSS02
Record Dates: First submitted 2019-07-10; First posted 2019-07-29 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Reference Standards

STUDY DESIGN:
Intervention Model Description: Healthy adult volunteers that meet inclusion/exclusion criteria will be randomized to receive 2 of the 4 products on bilateral site on the abdomen and/or groin.
Who Masked: Outcomes Assessor
Masking Description: Study products cannot be blinded to staff member(s) performing product applications, sample collections.
  Staff member(s) performing bacterial enumeration will be blinded from the identification of all study product assignments.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (4):
- Investigational Product (Experimental): Skin will be prepared with investigational product
  Interventions: Combination Product: Investigational Product
- Reference Standard (Other): Skin will be prepared with reference standard
  Interventions: Other: Reference Standard
- Active Control (Active Comparator): Skin will be prepared with active comparator
  Interventions: Combination Product: Active Comparator
- Negative Control (Other): Skin will be prepared with negative control
  Interventions: Other: Negative Control

INTERVENTIONS:
Combination Product: Investigational Product — 2%(w/v) Chlorhexidine in 70%(v/v) Isopropyl skin preparation
  Arms: Investigational Product
Other: Reference Standard — 60% (v/v) 1-propanol skin preparation
  Arms: Reference Standard
Combination Product: Active Comparator — ChloraPrep® SEPP® skin preparation
  Arms: Active Control
Other: Negative Control — 0.9% Normal Saline skin preparation
  Arms: Negative Control

SUMMARY:
This single site study is a randomized, controlled, partially-blinded design enrolling a minimum of 516 healthy volunteers, where each subject will receive two of the planned study products on the product application sites of the abdomen and/or groin.

DETAILED DESCRIPTION:
To demonstrate the antimicrobial activity of the Investigational Product (IP) by comparing counts of resident skin microbes, obtained after IP application to intact skin of the abdomen and groin, to counts obtained prior to application.

ELIGIBILITY:
Inclusion Criteria:

1. Read, understand, and provide signed informed consent.
2. Are healthy subjects in good general health
3. Are 18 years of age or older
4. If females of childbearing potential, are using an acceptable form of birth control for at least 28 days immediately preceding Day 1 and throughout the duration of the study. Acceptable methods are established, effective hormonal contraception (oral/implant/injectable/transdermal/intra-vaginal), intra-uterine device [IUD], diaphragm with spermicide, condom with spermicide, abstinence, bilateral tubal ligation, or are in a monogamous relationship with a partner who has had a vasectomy
5. In the case of females of childbearing potential, have a negative urine pregnancy test (UPT) on Product Application Day prior to any applications of the study products.
6. Are free of any systemic or dermatologic disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs.
7. Have minimal Screening Day bacterial count.

Exclusion Criteria:

1. Have had exposure to topical or systemic antimicrobials or any other product known to affect the normal microbial flora of the skin, antibiotics or steroids (other than hormones for contraception or post-menopausal reasons) within the product restriction period and for the remainder of the study. Restrictions include, but are not limited to antimicrobial soaps, antiperspirants/deodorants, shampoos, lotions, perfumes, after shaves, and colognes.
2. Subjects who have a history of skin allergies.
3. Have known allergies or sensitivity to vinyl, latex (rubber), alcohols, metals, inks, common consumer/beauty products, tape adhesives, or to common antibacterial agents found in soaps, lotions, or ointments, particularly chlorhexidine, or any other product components.
4. Swimming in chemically treated pools or bathing in hot tubs, spas and whirlpools within the product restriction period and for the remainder of the study.
5. Use of tanning beds, hot waxes, or depilatories, including shaving (in the applicable product application areas) within the product restriction period and for the remainder of the study.
6. Have had exposure of the product application sites to strong detergents, acids, bases, bug repellant, fabric softener-treated clothing, UV treated clothing, other household chemicals in the applicable product application areas or other irritants during the product restriction period or during the study period.
7. Have a history of skin cancer within 6 inches of applicable product application areas, or are currently being treated for skin cancer or have received treatment for any type of internal cancer within the 5 years prior to enrollment.
8. Subjects who have a history of asthma, diabetes, hepatitis B or C, an organ transplant, mitral valve prolapse with a heart murmur, congenital heart disease, lupus, Crohn's disease, medicated multiple sclerosis, internal prosthesis or any immunocompromised conditions (such as AIDS or HIV positive).
9. A currently active skin disease or inflammatory skin condition (for example contact dermatitis) anywhere on the body.
10. Any tattoos or scars (including stretch marks) on the product application sites or within 2 inches of the product application sites; skin blemishes or warts may be permissible with the specific approval of the Investigator or consulting physician.
11. Dermatoses, cuts, lesions, active skin rashes, scabs, breaks in the skin or other skin disorders within 6 inches on or around the product application sites.
12. Subjects who have showered or bathed within at least 72 hours of the Product Application Day. Sponge baths may be taken, however, the lower abdomen and upper thigh region must be avoided.
13. Subjects who have an irritation score of 1 or greater (any redness, swelling, rash, or dryness present at any product application area) for any individual skin condition prior to the Product Application Day baseline sample collection.
14. Are females who are pregnant, plan to become pregnant during the study, or are breastfeeding a child.
15. Are unable to adhere to or understand the protocol.
16. Have used an investigational drug or participated in an investigational study within 30 days prior to signing the informed consent for this study or are currently participating in a clinical study.
17. Are employed by or are a family member of staff of BD or the study site conducting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1935 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Evic Product Testing Romania S.R.L., Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only treated if screening day baseline bacterial counts met the inclusion criteria.
  Participants were treated with 2 out of 4 study products (Investigational Product, Reference Standard, Active control and Negative Control) 1 on the left side of the body (both groin and abdomen), 1 on the right side of the body (both groin and abdomen).
Groups:
- All Study Participants: Study Participants that were treated
Period: Overall Study
Arm/Group | All Study Participants
Started | 1121
Treated With Investigational Product | 609
Treated With Reference Standard | 419
Treated With Active Control | 609
Treated With Negative Control | 605
Completed | 1121
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All Participants Who Completed Evaluations
Arm/Group | All Study Participants
Number analyzed (Participants) | 1121
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205
  Male | 916
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1121
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1120
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Romania | 1121

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial log10 Reductions From Baseline for Investigational Product and Reference Standard at 30 Seconds and 6 Hours Post-product Application
Description: Bacterial log10/cm^2 reductions for abdominal and groin sites post-product application (30 seconds and 6 hours) using the Investigational Product or Reference Standard.
Time Frame: 30 seconds and 6 hours post-product application
Population: This outcome includes test requirements outlined by Health Canada (HC) for an investigational product to demonstrate immediate and persistent antimicrobial activity against a reference standard, 60% v/v 1-Propanol. This outcome does not include negative and active control comparators. Analysis only includes participants with required treatment day baseline bacterial counts at each anatomical site at baseline and non-missing data at 30 seconds and 6 hours post-product application.
Measure: Mean (95% Confidence Interval); unit: Log10 CFU/cm^2
Groups:
- Investigational Product: Single Swabstick impregnated with 1.75mL of 2%(w/v) chlorhexidine gluconate in 70%(v/v) isopropyl alcohol
- Reference Standard: 1.75 mL of 60% (v/v) 1-propanol applied with a single Swabstick
Arm/Group | Investigational Product | Reference Standard
Number analyzed (Participants) | 609 | 419
Log10 CFU/cm^2
  Abdomen 30 Seconds: number analyzed (Participants) | 291 | 207
  Abdomen 30 Seconds | 2.53 [2.39 to 2.67] | 2.70 [2.53 to 2.87]
  Abdomen 6 hours: number analyzed (Participants) | 291 | 207
  Abdomen 6 hours | 2.68 [2.54 to 2.82] | 2.73 [2.57 to 2.89]
  Groin 30 Seconds: number analyzed (Participants) | 295 | 198
  Groin 30 Seconds | 3.69 [3.53 to 3.84] | 4.07 [3.89 to 4.25]
  Groin 6 hours: number analyzed (Participants) | 295 | 198
  Groin 6 hours | 3.89 [3.73 to 4.04] | 4.08 [3.90 to 4.27]

2. Primary Outcome: Antimicrobial Activity (Efficacy): log10 CFU/cm2 of Resident Microbes on Skin at Baseline and 10 Minutes Post-product Application.
Description: Evaluation of antimicrobial activity will be based on log10 CFU/cm2 of resident microbes on skin before and after each product application on the abdomen and groin.
Time Frame: Baseline and 10 minutes post-product application
Population: This outcome includes FDA test requirements for an investigational product (IP) to demonstrate superior antimicrobial activity to a negative control and non-inferiority to an active control at the immediate time point of 10 minutes on the abdomen and groin. This outcome does not require a reference standard. Analysis only includes participants with required treatment day baseline bacterial counts at each anatomical site at baseline and non-missing data at 10 minutes post-product application.
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Groups:
- Active Control: ChloraPrep® SEPP® clear applicator- 2% (w/v) chlorhexidine gluconate in 70% (v/v) isopropyl alcohol
- Negative Control: 1.75mL 0.9% Normal saline applied with a single Swabstick
Arm/Group | Investigational Product | Active Control | Negative Control
Number analyzed (Participants) | 609 | 609 | 605
Log10 CFU/cm^2
  Abdomen Baseline: number analyzed (Participants) | 291 | 307 | 303
  Abdomen Baseline | 3.93 (.61) | 3.88 (.58) | 4.00 (.62)
  Abdomen 10 Minutes: number analyzed (Participants) | 291 | 307 | 303
  Abdomen 10 Minutes | 1.34 (1.13) | 1.31 (1.04) | 3.19 (.80)
  Groin Baseline: number analyzed (Participants) | 295 | 293 | 295
  Groin Baseline | 6.14 (.47) | 6.16 (.46) | 6.17 (.48)
  Groin 10 Minutes: number analyzed (Participants) | 295 | 293 | 295
  Groin 10 Minutes | 2.46 (1.36) | 2.70 (1.32) | 4.84 (.70)
Statistical Analysis 1: Comparison: Investigational Product vs Active Control; Abdomen at 10 minutes post-product application. Average treatment effect (ATE) of the Investigational Product compared to the Active Control on the abdomen at 10 minutes post-product application. ATE was calculated using a linear regression model for each body site used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — A non-inferiority criterion with a 0.5 log10 margin will be implemented for the average treatment effect (ATE) of the Investigational Product compared to the Active Control (i.e., the upper two-sided 95% confidence bound of the post-product application bacterial load corrected for pre-product application bacterial load of the Investigational Product - Active Control should be less than 0.5 log10); Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.15 to 0.16]
Statistical Analysis 2: Comparison: Investigational Product vs Active Control; Groin at 10 minutes post-product application. Average treatment effect (ATE) of the Investigational Product compared to the Active Control on the groin at 10 minutes post-product application. ATE was calculated using a linear regression model for each body site used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.43 to -0.05]
Statistical Analysis 3: Comparison: Investigational Product vs Negative Control; Abdomen at 10 minutes post-product application. Average treatment effect (ATE) of the Investigational Product compared to the Negative Control on the abdomen at 10 minutes post-product application. ATE was calculated using a linear regression model for each body site used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Superiority; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [1.66 to 1.97]
Statistical Analysis 4: Comparison: Investigational Product vs Negative Control; Groin at 10 minutes post-product application. Average treatment effect (ATE) of the Investigational Product compared to the Negative Control on the groin at 10 minutes post-product application. ATE was calculated using a linear regression model for each body site used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Superiority; Mean Difference (Final Values) = 2.38, 95% CI 2-sided [2.19 to 2.56]

3. Primary Outcome: Responder Rate at 6 Hours Post-Product Application on the Abdomen.
Description: Number of participants with bacterial reduction greater than or equal to baseline (0).
Time Frame: 6 hours post-product application
Population: This outcome includes FDA test requirements to demonstrate persistence of the investigational product (IP) at 6 hours post-product application on the abdomen. This outcome does not require a reference standard. Analysis only includes participants with required treatment day baseline bacterial counts on the abdomen at baseline and non-missing data at 6 hours post-product application.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Active Control | Negative Control
Number analyzed (Participants) | 291 | 307 | 303
Participants | 286 | 305 | 265

4. Primary Outcome: Responder Rate at 6 Hours Post-Product Application on the Groin.
Description: Number of participants with bacterial reduction greater than or equal to baseline (0).
Time Frame: 6 hours post-product application
Population: This outcome includes FDA test requirements to demonstrate persistence of the investigational product (IP) at 6 hours post-product application on the groin. This outcome does not require a reference standard. Analysis only includes participants with required treatment day baseline bacterial counts on the groin at baseline and non-missing data at 6 hours post-product application.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Active Control | Negative Control
Number analyzed (Participants) | 295 | 293 | 295
Participants | 295 | 293 | 291

5. Secondary Outcome: Antimicrobial Activity (Efficacy): log10 CFU/cm2 of Resident Microbes on Skin at Baseline and 30 Seconds Post-product Application.
Description: as for outcome 2
Time Frame: Baseline and 30 seconds post-product application
Population: This outcome includes FDA test requirements for an investigational product (IP) to demonstrate superior antimicrobial activity to a negative control and non-inferiority to an active control at the immediate time point of 30 seconds on the abdomen and groin. This outcome does not require a reference standard. Analysis only includes participants with required treatment day baseline bacterial counts at each anatomical site at baseline and non-missing data at 30 seconds post-product application.
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Arm/Group | Investigational Product | Active Control | Negative Control
Number analyzed (Participants) | 609 | 609 | 605
Log10 CFU/cm^2
  Abdomen Baseline: number analyzed (Participants) | 291 | 307 | 303
  Abdomen Baseline | 3.93 (.61) | 3.88 (.58) | 4.00 (.62)
  Abdomen 30 seconds: number analyzed (Participants) | 291 | 307 | 303
  Abdomen 30 seconds | 1.40 (1.19) | 1.30 (1.06) | 3.43 (.72)
  Groin Baseline: number analyzed (Participants) | 295 | 293 | 295
  Groin Baseline | 6.14 (.47) | 6.16 (.46) | 6.17 (.48)
  Groin 30 seconds: number analyzed (Participants) | 295 | 293 | 295
  Groin 30 seconds | 2.46 (1.36) | 2.80 (1.34) | 5.20 (.62)
Statistical Analysis 1: Comparison: Investigational Product vs Active Control; Abdomen at 30 seconds post-product application. Average treatment effect (ATE) of the Investigational Product compared to the Active Control on the abdomen at 30 seconds post-product application. ATE was calculated using a linear regression model for each body site used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.08 to 0.23]
Statistical Analysis 2: Comparison: Investigational Product vs Negative Control; Abdomen at 30 seconds post-product application. Average treatment effect (ATE) of the Investigational Product compared to the Negative Control on the abdomen at 30 seconds post-product application. ATE was calculated using a linear regression model for each body site used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Superiority; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [1.84 to 2.15]

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Investigational Product | Reference Standard | Active Control | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/609 | 0/419 | 0/609 | 0/605
Serious Adverse Events (participants affected / at risk) | 0/609 | 0/419 | 0/609 | 0/605
Other Adverse Events (participants affected / at risk) | 0/609 | 0/419 | 0/609 | 0/605

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT04035161/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT04035161/SAP_001.pdf